CLINICAL TRIAL: NCT04585152
Title: Randomized Controlled Trial Comparing Rituximab to Mycophenolate Mofetil in Children With Steroid-dependent Idiopathic Nephrotic Syndrome.
Brief Title: Rituximab Versus Mycophenolate Mofetil in Children With Steroid-dependent Idiopathic Nephrotic Syndrome.
Acronym: RTXvsMMF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Giannina Gaslini (Other)
Collaborators: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Gian Marco Ghiggeri MD, PhD, MD, director of Nephrology, Dialysis and Transplantation Unit, Istituto Giannina Gaslini
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTXvsMMF
Record Dates: First submitted 2020-09-16; First posted 2020-10-14 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Nephrotic Syndrome Steroid-Dependent
Keywords: nephrotic syndrome treatment; rituximab; Mycophenolate Mofetil
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Intervention Model Description: The RTX-MMF trial is an open-label, two-parallel-arm, controlled and randomized clinical trial testing the superiority of RTX over MMF in maintaining steroid free disease remission in patients with SDNS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab biosimilar (Experimental): Drug Name: Rituximab biosimilar monoclonal anti-CD20 antibody Why: Anti-body/antigen interaction results in cell apoptosis and reduced CD20 positive cell related activities (of note CD20 is mostly represented on B cells but also in Th17 cells) How: RTX IV: for dosage between 100 and 250 mg Rituximab will be diluted in 100 ml of normal saline and administered at 2 ml/h for the first 30'; 3 ml/h for the second 30'; 6 ml/h for the third 30'; 15 ml/h until the end. For dosage between 260 and 500 mg Rituximab will be diluted in 250 ml of normal saline and administered at 6 ml/h for the first 30'; 9 ml/h for the second 30'; 18 ml/h for the third 30'; 36 ml/h until the end. For dosage between 510 and 1000 mg Rituximab will be diluted in 500 ml of normal saline and administered at 9 ml/h for the first 30'; thereafter, the infusion rate can be doubled every 30 minutes up to a maximum of 72 ml/h.
  Where: in Hospital When and how much: once; diluted in 1000 ml of normal saline.
  Interventions: Drug: Rituximab Biosimilar
- Mycophenolate mofetil (Active Comparator): Drug Name: Mycophenolate Mofetil (MMF)
  Why: selective and reversible inhibition of inosine monophosphate dehydrogenase with inhibition that particularly affects lymphocytes since they rely almost exclusively de novo purine synthesis Procedures: MMF 1,200 mg/m2 orally divided in 2 daily doses
  Interventions: Drug: Rituximab Biosimilar

INTERVENTIONS:
Drug: Rituximab Biosimilar — for dosage between 100 and 250 mg Rituximab will be diluted in 100 ml of normal saline and administered at 2 ml/h for the first 30'; 3 ml/h for the second 30'; 6 ml/h for the third 30'; 15 ml/h until the end. For dosage between 260 and 500 mg Rituximab will be diluted in 250 ml of normal saline and administered at 6 ml/h for the first 30'; 9 ml/h for the second 30'; 18 ml/h for the third 30'; 36 ml/h until the end. For dosage between 510 and 1000 mg Rituximab will be diluted in 500 ml of normal saline and administered at 9 ml/h for the first 30'; thereafter, the infusion rate can be doubled every 30 minutes up to a maximum of 72 ml/h.

SUMMARY:
Anti-CD20 monoclonal antibodies are emerging as the steroid-sparing therapy of choice for nephrotic syndrome.This Randomized Clinical Trial seeks to evaluate whether Rituximab biosimilar maintains drug-free disease remission in patients with steroid-dependent nephrotic syndrome for 12-24 months and verify its superiority vs. mycophenolate mofetil (1,200 mg/m2 orally in 2 daily doses). The investigators will compare the risk of relapse to test this hypothesis (primary outcome). Secondary objectives will include assessing short- and long-term side-effects and developing specific biomarkers of sensitivity to therapy. Patients will be recruited, treated and followed at IRCCS G Gaslini and IRCCS Bambino Gesù where laboratory studies will be performed at in-site facilities.

DETAILED DESCRIPTION:
Idiopathic nephrotic syndrome (NS) is a podocyte renal disease characterized by loss of the impermeability functions versus circulating proteins, causing severe proteinuria and hypo-albuminaemia with edema. According to 2019 KDIGO guidelines administration of low-dose prednisone is suggested to maintain remission in SDNS (steroid dependant nephrotic syndrome), and mycophenolate mofetile (MMF) or calcineurin inhibitors (CNI) or Rituximab as corticosteroid-sparing agents for children who develop serious corticosteroid-related adverse effects. Given the toxicity of cyclophosphamide and CNI in long-term administration, there is the need to clarify which is, between MMF and rituximab, the most effective approach.

The RTX vs MMF trial is an open-label, two-parallel-arm, controlled and randomized clinical trial testing the superiority of RTX over MMF (1,200 mg/m2 orally in two daily doses) in maintaining steroid free disease remission in patients with SDNS.

Eligible participants are children and young adults (age between 3 and 24 years) with nephrotic syndrome who are dependent on prednisone 0.3-1mg/Kg/day and have received prednisone for at least six months before enrolment. Previous treatment with MMF will be allowed. All participants will enter a 45 days run-in period, during which children treated with steroids alone will start MMF and will taper steroids after 15 days by 0.3 mg/kg per week until complete withdrawal. Patients already receiving MMF alone will continue the treatment. During the same period, instruction on urine collection and dipstick readings will be carefully reviewed and compliance assessed. After run-in period, children will be randomized to either the intervention arm (Rituximab, 375 mg/m2) or the comparator arm (continuing or starting MMF). In the intervention arm, 1 month after infusion MMF will be decreased by 50% and withdrawn within 2 additional weeks, whereas MMF will be maintained in the comparator. All patients will be followed for up to 24 months. In case of relapses during this period (see outcome section for definition) patients will be treated with oral prednisone (60 mg/sqm day). Following remission, steroids will be maintained at the initial dose for 7 days and then tapered off by 0.3 mg/kg per week until complete withdrawal in patients of the MMF arm. Patients of the intervention arm will instead be treated with another infusion of RTX (same dose) immediately following steroid-induced remission. After infusion of RTX, steroids will be maintained at the initial dose for 7 days and then tapered off by 0.3 mg/kg per week until complete withdrawal. In this way relapsed patients in both arms will receive the same cumulative dose of prednisone. In case following relapse of proteinuria patients fail to respond to prednisone (they will terminate the study and be considered as treatment failure). The study allows drop-in from one arm to the other after 2 relapses (i.e., investigators will be allowed to use RTX in the comparator arm and vice versa MMF in intervention arm). The economic balance will be calculated on the basis of RTX doses needed to maintain remittance.

All patients will be followed for 24 months. In person visits will occur at enrollment, at T0 (infusion), after 1 month and every 3/6 months later.

The investigators are going to enroll 160 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 and 24 years
* Prednison dependent steroid syndrome 0.3-1mg/Kg/day and receive prednisone for at least six months before enrolment. Steroid dependence is defined by two consecutive relapse during corticosteroid therapy or within 14 days of ceasing therapy.
* Ability to provide consent and assent: parents'/guardian's written informed consent, and child's assent given before any study-related procedure not part of the subject's normal medical care, with the understanding that consent may be withdrawn by the subject any time without prejudice to his or her future medical care.

Exclusion Criteria:

* Positivity to autoimmunity tests (ANA, nDNA, ANCA)
* Reduction of C3 levels.
* eGFR<90/ml/min/1,73 m2 valuated according to revised Bedside Schwartz Formula for patients between 2 and 17 years and with CKD-EPI Creatinine 2009 Equation for 18 years old patients.
* Pregnancy
* Neoplasm
* Infections: previous or actual HBV (with HBeAb positivity) or HCV infection CD20 B lymphocytes count <2,5%
* Treatment with Rituximab in the last 6 months

Ages: 3 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Comparison between RTX and MMF, considering remission intervals (in months) in the two cohorts | 12-24 months
  Comparison between RTX and MMF to maintain remission of NS for 12-24 months in children with primary SDNS. All the participats (n=160) will document their proteinuria and their urine will be analyzed periodically (at least every three months); relapse is defined by uPCR ≥2000 mg/g (≥ 200 mg/mmol) or > 3+ protein on urine dipstick for 3 consecutive days (KDIGO Clinical Practice Guideline for Glomerulonephritis, Kidney International Supplement, 2012 2, 163-171) and complete remission is defined by uPCR <200 mg/g (<20 mg/mmol) or o1+ of protein on urine dipstick for 3 consecutive days (KDIGO Clinical Practice Guideline for Glomerulonephritis, Kidney International Supplement, 2012 2, 163-171).

SECONDARY OUTCOMES:
RTX safety by evaluation and documentation of side effects measuring frequency and severity of any treatment-related adverse events as assessed by CTCAE v4.0 | 36 months
  A second result of the study will be based on the side-effects that RTX may induce: the investigators will record and measure frequency and severity of any treatment-related adverse events as assessed by CTCAE v4.0

OTHER OUTCOMES:
Biomarkers of immune competence: mononuclear cells (PBMCs) by cytometry, serum immunoglobulin | 36 months
  Identification of biomarkers of response to RTX and immune competence in patients treated with RTX vs. patients treated with MMF.
  Mononuclear cells (PBMCs) will be characterized by flow cytometry to investigate any difference between the two arms. Samples for cell analysis will be obtained at time 0 and after 3, 12 and 24 months; the same analysis will be performed in case of relapse. In parallel, total IgG, IgA and IgM levels will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: GianMarco Ghiggeri, MD, Principal Investigator — Istituto Giannina Gaslini
Locations (1):
- IRCCS G. Gaslini, Genova, Italy

IPD SHARING:
Plan to Share IPD: Yes
Yes The completed study will be summarized in a final report that accurately and completely presents the study objectives, methods, results, limitations of the study, and interpretation of findings.
  The first publication will be an in extenso publication of the results of the validation of the project.
  The Authors of this study protocol will inform the contributing investigators in advance about any plans to publish or present data from this randomized controlled clinical trial. Any publications and presentations of the results (abstract in journals or newspapers, oral presentations, etc.), either in whole or in part, by Investigators or their representatives will require pre-submission review by the Authors of this study protocol.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: it will be public on peer reviewed journal
Access Criteria: it will be public on peer reviewed journal

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526
- [Derived] Lugani F, Angeletti A, Ravani P, Vivarelli M, Colucci M, Caridi G, Verrina E, Emma F, Ghiggeri GM. Randomised controlled trial comparing rituximab to mycophenolate mofetil in children and young adults with steroid-dependent idiopathic nephrotic syndrome: study protocol. BMJ Open. 2021 Nov 29;11(11):e052450. doi: 10.1136/bmjopen-2021-052450. PMID 34845071